CLINICAL TRIAL: NCT00926471
Title: A Cognitive-Behavioral Intervention for Children With Autism Spectrum Disorders
Brief Title: Social Skills and Anxiety Reduction Treatment for Children and Adolescents With Autism Spectrum Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susan White, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K01MH079945 (NIH); K01MH079945 (NIH); DDTR B2-MBA
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Autistic Disorder; Child Development Disorders, Pervasive
Keywords: Autism; Anxiety; Autism Spectrum Disorders with Comorbid Anxiety
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (CBT) Program (Experimental): Participants will receive a treatment program involving CBT plus adjunctive group counseling and parent training.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT) Program
- Wait list control (No Intervention): Participants will be placed on a 12-week wait list with no active treatment

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) Program — 12 to 14 weekly sessions of individual CBT and parent training with 5 sessions of group counseling every other week
  Arms: Cognitive Behavioral Therapy (CBT) Program

SUMMARY:
This study will develop and test a treatment aimed at reducing anxiety in social situations for children and adolescents with autism spectrum disorders.

DETAILED DESCRIPTION:
Autism spectrum disorders (ASDs) are developmental disorders with similar features, including problems communicating, problems interacting socially, and the presence of routines or repetitive behaviors. These disorders can have a range of severities. They include autistic disorder, Asperger's syndrome, and pervasive developmental disorder not otherwise specified (PDD-NOS). In addition to their core impairment in social functioning, children and adolescents with ASDs often have anxiety about social interactions, which compounds their difficulties and can limit the benefits of treatment. This study will develop and test a treatment program for developing social skills and reducing anxiety in children and adolescents with ASDs.

Participation in this study will last 12 to 14 weeks, with follow-up visits occurring 3 and 12 months after that. Participants will be randomly assigned to receive the treatment program either immediately or after being on a wait list. The treatment program will consist of 12 to 14 weekly individual therapy sessions that teach children and adolescents about ASDs, use cognitive-behavioral interventions to address problematic thinking and acting, deliver social skills instruction, and give opportunities to practice skills-including some practice outside the clinic in naturalistic settings. Every 2 weeks, starting at Week 4, children and adolescents will also attend group sessions to discuss strategies and practice social skills. Parents of the participants will be included at the end of each individual session for several minutes. After the participants assigned to immediate treatment complete the program, participants from the wait list will be offered the treatment.

Child and adolescent participants and their parents will complete assessments at baseline, midpoint in treatment, post-treatment (Week 12 or 14), and 3- and 12-month follow-ups. Participants assigned to the wait list condition will complete assessments only at baseline, before entering treatment (Week 12 or 14), and after completing treatment. Assessments will involve questionnaires about social and emotional functioning, interviews with study researchers, and surveys on satisfaction with the study. The child or adolescent's primary teacher will also complete questionnaires about the child.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism, Asperger's syndrome, or pervasive developmental disorders not otherwise specified (PDD-NOS), as determined by clinical interview and supported by the Autism Diagnostic Interview-Revised (ADI-R) and Autism Diagnostic Observation Schedule (ADOS)
* Has completed assessment of brief verbal intelligence quotient (IQ), with a score of 70 or higher on the Weschler Abbreviated Scale of Intelligence (WASI)
* Symptoms of anxiety, defined as a clinical severity rating of 4 or higher on one of the following sections of the Anxiety Disorders Interview Schedule for Children (ADIS-C) and parents (ADIS-P): generalized anxiety disorder (GAD), social phobia, specific phobia, agoraphobia, or separation anxiety disorder
* If on psychiatric medication, on stable dose for 4 weeks prior to baseline assessment with no planned changes to medication for anxiety

Exclusion Criteria:

* Psychopathology that warrants a different type of immediate clinical care
* Severe aggression, as determined by clinical judgment
* Mental retardation, as reported by parents or in previous psychoeducational testing supplied by parents
* Child and family currently in therapy

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Child and Adolescent Symptom Inventory 20-Item Anxiety Subscale (CASI-20) | Measured at baseline, post-treatment, and 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Susan W White, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Polytechnic Institute and State University, Blacksburg, Virginia, United States